CLINICAL TRIAL: NCT03412682
Title: A Phase 3, Multi-centre, Randomised, Double-blind, Active-controlled, Parallel-group Trial Investigating the Efficacy and Safety of FE 999315 Following 8 Weeks of Treatment for Mild to Moderate Active Ulcerative Colitis in Japanese Subjects
Brief Title: To Evaluate the Efficacy and Safety of FE 999315 in Japanese Subjects With Mild to Moderate Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000234
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative colitis; FE999315; Mesalazine; Colitis; Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — Budesonide; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Budesonide (6 mg) (Experimental)
  Interventions: Drug: Budesonide (6 mg)
- Budesonide (9 mg) (Experimental)
  Interventions: Drug: Budesonide (9 mg)
- Mesalazine (3,600 mg) (Active Comparator)
  Interventions: Drug: Mesalazine (3,600 mg)

INTERVENTIONS:
Drug: Budesonide (6 mg) — Budesonide (6 mg) administered once a day along with three mesalazine placebo three times a day, over an 8-week treatment period.
  Other Names: FE 999315
  Arms: Budesonide (6 mg)
Drug: Budesonide (9 mg) — Budesonide (9 mg) administered once a day along with three mesalazine placebo three times a day, over an 8-week treatment period.
  Other Names: FE 999315
  Arms: Budesonide (9 mg)
Drug: Mesalazine (3,600 mg) — Mesalazine (3,600 mg) administered once a day plus three mesalazine 400 mg three times a day, over an 8-week treatment period.
  Arms: Mesalazine (3,600 mg)

SUMMARY:
To demonstrate non-inferiority in efficacy of FE 999315 to mesalazine in patients with mild to moderate active ulcerative colitis after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 16 to 75 years old, diagnosed with ulcerative colitis.
* Diagnosis of ulcerative colitis in active phase of mild to moderate entity.
* Female patients must fulfill at least one of the following criteria: Post-menopausal (women ≥45 years with no menstrual period for at least 12 months without an alternative medical cause), surgically sterile, using a medically approved contraception throughout the trial period or her male partner using medically approved contraception throughout the trial period.
* Male patients must agree to use medically approved contraception throughout the trial period.

Exclusion Criteria:

* Patients with limited distal proctitis.
* Patients with infectious colitis.
* Patients with history of colectomy.
* Patients with severe diseases in other organs and systems.
* Evidence or history of toxic megacolon.
* Women who wish to become pregnant during the trial period

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline of total Ulcerative Colitis Disease Activity Index (UCDAI) scores after 8 weeks of treatment using the mucosal appearance score | After 8 weeks
  UCDAI is a four-component scale, used to determine the severity of ulcerative colitis. The four components assessed are stool frequency, rectal bleeding, mucosal appearance and physician's rating of disease activity. Score for each component can range between 0-3 and thus, the maximum overall score can be between 0-12. Higher score implies higher disease severity.

SECONDARY OUTCOMES:
Percentage of subjects achieving clinical remission after 8 weeks of treatment | 8 weeks
Percentage of subjects achieving 0 score for subscores of rectal bleeding, stool frequency and mucosal appearance (normal mucosa) in UCDAI after 8 weeks of treatment | 8 weeks
Percentage of subjects achieving clinical improvement after 8 weeks of treatment | 8 weeks
Percentage of subjects achieving endoscopic improvement after 8 weeks of treatment for subjects with baseline UCDAI mucosal appearance subscore greater than equal to [≥]1 | 8 weeks
Percentage of subjects achieving symptom resolution after 2 weeks of treatment | 2 weeks
Percentage of subjects achieving symptom resolution after 4 weeks of treatment | 4 weeks
Percentage of subjects achieving symptom resolution after 8 weeks of treatment | 8 weeks
Percentage of subjects with endoscopic healing after 8 weeks of treatment | 8 weeks
Change from baseline in partial UCDAI score at 2 weeks | 2 weeks
Change from baseline in partial UCDAI score at 4 weeks | 4 weeks
Change from baseline in partial UCDAI score at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (72):
- Japan (72):
  - Ferring Investigator Site JPN27, Nagoya, Aichi-ken
  - Ferring Investigator Site JPN52, Toyoake-shi, Aichi-ken
  - Ferring Investigator Site JPN47, Toyota-shi, Aichi-ken
  - Ferring Investigator Site JPN69, Abiko-shi, Chiba
  - Ferring Investigator Site JPN68, Kashiwa-shi, Chiba
  - Ferring Investigator Site JPN53, Urayasu-shi, Chiba
  - Ferring Investigator Site JPN08, Matsuyama, Ehime
  - Ferring Investigator Site JPN50, Fukui-shi, Fukui
  - Ferring Investigator Site JPN51, Chikushino-shi, Fukuoka
  - Ferring Investigator Site JPN31, Fukuoka, Fukuoka
  - Ferring Investigator Site JPN64, Fukuoka, Fukuoka
  - Ferring Investigator Site JPN28, Kitakyushu, Fukuoka
  - Ferring Investigator Site JPN19, Kitakyushu-shi, Fukuoka
  - Ferring Investigator Site JPN23, Kitakyushu-shi, Fukuoka
  - Ferring Investigator Site JPN35, Kitakyushu-shi, Fukuoka
  - Ferring Investigator Site JPN38, Kurume-shi, Fukuoka
  - Ferring Investigator Site JPN36, Gifu, Gifu
  - Ferring Investigator Site JPN17, Takasaki-shi, Gunma
  - Ferring Investigator Site JPN46, Hatsukaichi, Hiroshima
  - Ferring Investigator Site JPN11, Asahikawa-shi, Hokkaido
  - Ferring Investigator Site JPN59, Hakodate-shi, Hokkaido
  - Ferring Investigator Site JPN61, Sapporo, Hokkaido
  - Ferring Investigator Site JPN14, Kobe, Hyōgo
  - Ferring Investigator Site JPN13, Nishinomiya-shi, Hyōgo
  - Ferring Investigator Site JPN40, Nishinomiya-shi, Hyōgo
  - Ferring Investigator Site JPN43, Kasama-shi, Ibaraki
  - Ferring Investigator Site JPN24, Koga-shi, Ibaraki
  - Ferring Investigator Site JPN22, Tsuchiura-shi, Ibaraki
  - Ferring Investigator Site JPN41, Takamatsu, Kagawa-ken
  - Ferring Investigator Site JPN02, Kagoshima, Kagoshima-ken
  - Ferring Investigator Site JPN29, Kagoshima, Kagoshima-ken
  - Ferring Investigator site JPN05, Yokohama, Kanagawa
  - Ferring Investigator Site JPN33, Yokohama, Kanagawa
  - Ferring Investigator Site JPN67, Yokohama, Kanagawa
  - Ferring Investigator Site JPN63, Nankoku-shi, Kochi
  - Ferring Investigator Site JPN34, Kyoto, Kyoto
  - Ferring Investigator Site JPN48, Tsu, Mie-ken
  - Ferring Investigator Site JPN12, Yokkaichi-shi, Mie-ken
  - Ferring Investigator site JPN04, Sendai, Miyagi
  - Ferring Investigator Site JPN44, Nagasaki, Nagasaki
  - Ferring Investigator Site JPN66, Nagasaki, Nagasaki
  - Ferring Investigator Site JPN62, Kashihara-shi, Nara
  - Ferring Investigator Site JPN55, Niigata, Niigata
  - Ferring Investigator Site JPN37, Beppu-shi, Oita Prefecture
  - Ferring Investigator Site JPN01, Ōita, Oita Prefecture
  - Ferring Investigator Site JPN72, Ōita, Oita Prefecture
  - Ferring Investigator Site JPN65, Okayama, Okayama-ken
  - Ferring Investigator site JPN07, Fujiidera-shi, Osaka
  - Ferring Investigator Site JPN10, Osaka, Osaka
  - Ferring Investigator Site JPN26, Osaka, Osaka
  - Ferring Investigator Site JPN30, Osaka, Osaka
  - Ferring Investigator Site JPN60, Sakai-shi, Osaka
  - Ferring Investigator Site JPN39, Suita-shi, Osaka
  - Ferring Investigator Site JPN21, Takatsuki-shi, Osaka
  - Ferring Investigator Site JPN57, Toyonaka-shi, Osaka
  - Ferring Investigator Site JPN03, Saitama-shi, Saitama
  - Ferring Investigator Site JPN09, Saitama-shi, Saitama
  - Ferring Investigator Site JPN49, Sakura-shi, Saitama
  - Ferring Investigator Site JPN42, Tokorozawa-shi, Saitama
  - Ferring Investigator Site JPN56, Tokorozawa-shi, Saitama
  - Ferring Investigator Site JPN70, Mibu, Tochigi
  - Ferring Investigator Site JPN32, Fuchū-shi, Tokyo
  - Ferring Investigator Site JPN20, Kodaira-shi, Tokyo
  - Ferring Investigator Site JPN15, Machida-shi, Tokyo
  - Ferring Investigator site JPN06, Meguro-ku, Tokyo
  - Ferring Investigator Site JPN58, Minato-ku, Tokyo
  - Ferring Investigator Site JPN71, Mitaka-shi, Tokyo
  - Ferring Investigator Site JPN18, Oume-shi, Tokyo
  - Ferring Investigator Site JPN54, Shinagawa-Ku, Tokyo
  - Ferring Investigator Site JPN45, Shinjuku-Ku, Tokyo
  - Ferring Investigator Site JPN16, Kofu, Yamanashi
  - Ferring Investigator Site JPN25, Hiroshima-shi, Hiroshima